CLINICAL TRIAL: NCT06847438
Title: Tailored Electronic Intervention to Improve Therapy in a Diverse Cohort of Patients With Heart Failure
Acronym: TAILORD-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Neal Dickert, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00006716
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Clinics will be randomly assigned to implement the checklist or to not implement the checklist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Optimized version of the EPIC-HF Checklist (Other): Patients of clinics that are randomized to implement the checklist will be sent the checklist in advance of their visit via their electronic medical record (EMR) portal.
  Interventions: Behavioral: Optimized version of the EPIC-HF Checklist
- EPIC-HF Checklist for Patients and Clinician-facing Decision Support (Other): Patients of clinics that are randomized to implement the checklist will be sent the checklist in advance of their visit via their electronic medical record (EMR) portal. During this period of the study, clinicians in intervention clinics will also have access to analogous decision-support via EMR.
  Interventions: Behavioral: Optimized version of the EPIC-HF Checklist; Behavioral: Clinician-facing Decision Support
- Standard of Care (Active Comparator): Patients of clinics that are randomized to the standard of care will not have the EPIC-HF checklist available for viewing in their electronic medical record (EMR).
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Optimized version of the EPIC-HF Checklist — The EPIC-HF checklist is a 1-page patient activation tool that contains approved and guideline-recommended medications and target doses for HFrEF. The EPIC-HF checklist allows patients to see recommended doses and categories of GDMT, which they can compare to their current medications and dosing. The EPIC-HF checklist has been refined and updated to include GDMT prescription and has been optimized for delivery through electronic medical record (EMR) systems. The checklist is being used as a patient activation/ discussion tool only and data entered on the checklist will not be collected for purposes of this study.
  Arms: EPIC-HF Checklist for Patients and Clinician-facing Decision Support; Optimized version of the EPIC-HF Checklist
Behavioral: Clinician-facing Decision Support — Information regarding GDMT (including target doses and medications) analogous to what is contained in the checklist will be provided to clinicians in intervention clinics. This information will be visible at the time of the encounter.
  Arms: EPIC-HF Checklist for Patients and Clinician-facing Decision Support
Behavioral: Standard of Care — Patients of clinics that are not implementing EPIC-HF checklist will not have the checklist available to them through the electronic medical record (EMR).
  Arms: Standard of Care

SUMMARY:
Recent medical guidelines for the management of heart failure (HF) have established a combination of specific classes of medications as the best treatment for patients with heart failure with reduced ejection fraction (HFrEF). However, studies have shown that these medications, known together as guideline-directed medical therapy (GDMT), are not being used in clinical practice less often than they could be. Several tools to promote broader use of these treatments (including patient checklists) have shown promise for increasing use of GDMT. However, these tools have not been broadly implemented within large health systems. The goal of this study is to see if using these tools broadly within cardiology clinics will increase the use of GDMT. This study is important because it could help improve the use of GDMT, which may lead to improved patient care and outcomes.

DETAILED DESCRIPTION:
The 2022 American College of Cardiology Foundation (ACCF)/American Heart Association (AHA)/Heart Failure Society of America (HFSA) and 2021 European Society of Cardiology (ESC) guidelines for the management of heart failure (HF) firmly establish that quadruple therapy with angiotensin receptor neprilysin inhibitors (ARNI), sodium glucose cotransporter-2 inhibitors (SGLT2i), evidence-based β-blockers, and mineralocorticoid receptor antagonists now form the foundational standard for guideline-directed medical therapy (GDMT) for patients with heart failure with reduced ejection fraction (HFrEF). Despite multiple randomized controlled trials establishing the clinical benefit of novel therapies like ARNI and SGLT2i, adoption of these novel therapeutic agents in clinical practice has been slower than expected. For example, a recent population-level cohort study using IQVIA Inc. National Prescription Audit data in the US showed that only 13.8% of patients with HFrEF were using sacubitril-valsartan from 2016-2019. Similarly, a recent retrospective cohort analysis of commercially insured patients with type 2 diabetes in the US demonstrated that only 8.7% were treated with an SGLT2i from 2015 to 2019. There is a need for interventions that increase utilization of these important medications.

The investigators have previously demonstrated a high burden of HF and suboptimal use of GDMT among a broad cohort of patients. There is a need to improve prescription of GDMT and to improve clinical outcomes for patients with HF with the use of evidence-based methods to improve care quality.

The EPIC-HF checklist is a patient activation tool that allows patients to see recommended doses and categories of GDMT, which they can use to compare to their current medications and dosing. In this implementation study, eight cardiology and heart failure clinics will be randomized to implement the EPIC-HF checklist or to perform standard of care for two 6-month periods. During the first 6-month period, patients will be provided with the EPIC-HF checklist prior to their clinic appointment via EMR message. During the second 6-month period, clinician-facing decision support for GDMT intensification will be added.

ELIGIBILITY:
Inclusion Criteria:

* Ejection fraction (EF) less than or equal to 40% by echocardiogram performed in the prior 18 months
* Diagnosis of heart failure

Exclusion Criteria:

* Heart failure (HF) etiology for which GDMT is not indicated: including hypertrophic or restrictive cardiomyopathy (e.g. amyloid cardiomyopathy), constrictive pericarditis, or complex congenital heart disease
* End-stage HF requiring continuous inotrope infusion, heart transplant, or left ventricular assist device
* Estimated glomerular filtration rate (eGFR) < 15 mL/min/1.73m^2
* Any conditions other than HF that are likely to alter the patient's status over 6 months, indicated by active hospice status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with GDMT Initiation or Intensification | 30 Days after Clinic Visit
  Changes in medication are assessed as the initiation or intensification of recommended heart failure medications including foundational GDMTs (angiotensin-converting enzyme inhibitors (ACEI)/angiotensin receptor blockers (ARB)/angiotensin receptor neprilysin inhibitors (ARNI), beta-blockers (BB), mineralocorticoid receptor antagonists (MRA), and sodium glucose cotransporter-2 inhibitors (SGLT2i)) as well as other guideline recommended therapies for HFrEF including ivabradine, digoxin, and soluble guanylate cyclase stimulators.

CONTACTS AND LOCATIONS:
Overall Officials: Neal W Dickert, MD, PhD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified participant data that underlie the results reported will be made available for sharing with other researchers.
Supporting Information: Study Protocol
Time Frame: Individual participant data will be available for sharing beginning 9 months after publication and 36 months following article publication.
Access Criteria: Data will be available for sharing with researchers who provide a methodologically sound proposal, in order to achieve the aims of the proposal. Proposals should be directed to njr@emory.edu. To gain access, requestors will need to sign a data access agreement.